CLINICAL TRIAL: NCT06844175
Title: A Prospective, Multicenter Cohort Study of Multidimensional Screening and Triple Drug Intervention in Young Patients with Chronic Obstructive Pulmonary Disease and Pre-chronic Obstructive Pulmonary Disease
Brief Title: Early Screening of Young COPD and Pre-COPD
Status: Not yet recruiting | Type: Observational
Sponsor: yanmengkang (Other)
Responsible Party: Sponsor-Investigator, yanmengkang, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: yanmeng kang
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (4):
- early COPD with placebo: 1. Age <50 years of age with at least 10 pack-years of smoking history and one of the following: FEV1/FVC< 0.7, abnormal computer tomography (CT) and a decline in FEV1 of at least 60mL/ year.
  2. Treatment with Placebo
- early COPD with triple inhalation therapy: 1. Age <50 years of age with at least 10 pack-years of smoking history and one of the following: FEV1/FVC< 0.7, abnormal computer tomography (CT) and a decline in FEV1 of at least 60mL/ year.
  2. Treatment with triple inhalation therapy
  Interventions: Drug: Budesonide, Glycopyrronium Bromide and Formoterol Fumarate Inhalation Aerosol
- pre-COPD with placebo: 1. It involved individuals of any age who had respiratory symptoms with or without structural (imaging-suggested emphysema) and/or functional abnormalities, without airflow limitation (FEV1/FVC≥0.70), and who may develop persistent airflow limitation over time.
  2. Treatment with Placebo
- pre-COPD with triple inhalation therapy: 1. It involved individuals of any age who had respiratory symptoms with or without structural (imaging-suggested emphysema) and/or functional abnormalities, without airflow limitation (FEV1/FVC≥0.70), and who may develop persistent airflow limitation over time.
  2. Treatment with triple inhalation therapy
  Interventions: Drug: Budesonide, Glycopyrronium Bromide and Formoterol Fumarate Inhalation Aerosol

INTERVENTIONS:
Drug: Budesonide, Glycopyrronium Bromide and Formoterol Fumarate Inhalation Aerosol — The intervention group was given budigfovir once a day, the dose was 160ug/7.2ug/4.8ug by inhalation
  Other Names: placebo
  Groups: early COPD with triple inhalation therapy; pre-COPD with triple inhalation therapy

SUMMARY:
At present, patients with early COPD and pre-COPD have not been paid attention to in clinical work. This study aims to actively screen such patients in high-risk groups to clarify their prevalence, monitor and analyze relevant clinical and biological indicators, and find sensitive indicators to assist in early diagnosis. Based on the updated definition of COPD in GOLD2022, we pay attention to the concept of early COPD and pre-COPD. After the completion of patient enrollment and data collection, we will further explore the effect of triple inhaled drug intervention on the development of lung function in patients with early COPD and pre-COPD, so as to provide clinical support for early screening and early treatment of COPD.

1. Patients with early COPD and pre-COPD were selected from 20 hospitals in 17 cities of Shandong province to understand the prevalence and basic characteristics of such diseases in the province, and then were divided into groups and treated.
2. The specificity and sensitivity of pulmonary function parameters (FEV1%,FEV1/FVC, DLco, etc.) and imaging parameters (MLD, Perc15, %LAA-950HU, etc.) alone or in combination in the diagnosis of early COPD and pre-COPD, and the predictive diagnostic model/system was established.
3. Treatment of early COPD and pre-COPD: eligible patients were given triple inhalation therapy or placebo, and the effects of triple inhalation therapy or not on clinical symptoms, pulmonary function, and imaging parameters were compared.

This study aims to determine the prevalence of early COPD in Shandong province and provide a reference for the treatment of this population.

DETAILED DESCRIPTION:
1. Basic information and related definitions: The basic information included age, gender, body mass index (BMI), smoking status (smoking index, passive smoking), biomass exposure, occupational exposure history of dust/gas/smoke, and family history of respiratory diseases. Participants' smoking status was categorized as never smoked, former smoker, or current smoker. Never smoked was defined as having smoked fewer than 100 cigarettes in the past. Current smoking was defined as baseline smoking. Previous smoking was defined as having smoked more than 100 cigarettes previously but not smoking for at least 6 months before baseline. The smoking index was defined as the number of packs of cigarettes smoked per day multiplied by the number of years smoked. Passive smoking was defined as smoke inhalation by non-smokers living with smokers for more than 1 year. Biomass exposure was defined as the use of biomass such as wood, crop residue, charcoal, grass, and manure for more than 1 year. Exposure to occupational dust/gas/smoke was defined as occupational exposure to dust/gas/smoke for more than 1 year during the lifetime of the subject. Family history of respiratory disease was defined as respiratory disease in parents, siblings, and childhood (e.g., chronic bronchitis, emphysema, asthma, COPD, cor pulmonalis, bronchiectasis, lung cancer, interstitial lung disease, obstructive sleep apnea-hypopnea syndrome) and a further visit to assess medication use history. Clinical symptoms included cough, expectoration, shortness of breath after exercise, suffocating wheezing, and dyspnea. Clinical symptoms were defined as the above symptoms not caused by other clear causes, and the cumulative time was not less than 2 months per year.
2. Questionnaire scores: ① Modified dyspnea scale (mMRC) : mainly used to evaluate the degree of dyspnea in COPD patients. The scale ranges from 0 to 4, with higher grades indicating more severe dyspnea, with grades 1 and 2 indicating "mild-to-moderate dyspnea," and grades 3 and 4 indicating "severe to very severe dyspnea. ②CAT score: a total of 8 questions covering symptoms, activities and conditions. Each question corresponds to a 0-5 point option on a 40-point scale, with higher scores indicating worse health status.
3. Pulmonary function: it was determined that the enrolled patients should stop using drugs that affect the test results and avoid related influencing factors before bronchodilation. Professional staff guided the patients to carry out respiratory training, and completed pulmonary ventilation and diffusion function tests. Ventilatory function was measured before and 15 minutes after inhalation of a bronchodilator (albuterol). forced vital capacity (FVC) and its percentage of predicted value (FVC%pred), forced expiratory volume in one second (FEV1) were recorded accurately. FEV1) and its percentage of predicted value (FEV1%pred), FEV1/FVC, maximum minute ventilation volume (MVV) and its percentage of predicted value (MVV%pred). The maximum midexpiratory flow (MMEF) was calculated. Diffusion capacity (DLCO) was measured by taking four to five quiet breaths in a single breath, then exhaling deeply to RV position, inhaling quickly to TLC position, holding breath for 10 seconds, and exhaling all the gas to RV position.

(3) Pulmonary function: it was determined that the enrolled patients should stop using drugs that affect the test results and avoid related influencing factors before bronchodilation. Professional staff guided the patients to carry out respiratory training, and completed pulmonary ventilation and diffusion function tests. Ventilatory function was measured before and 15 minutes after inhalation of a bronchodilator (albuterol). forced vital capacity (FVC) and its percentage of predicted value (FVC%pred), forced expiratory volume in one second (FEV1) were recorded accurately. FEV1) and its percentage of predicted value (FEV1%pred), FEV1/FVC, maximum minute ventilation volume (MVV) and its percentage of predicted value (MVV%pred). The maximum midexpiratory flow (MMEF) was calculated. Diffusion capacity (DLCO) was measured by taking four to five quiet breaths in a single breath, then exhaling deeply to RV position, inhaling quickly to TLC position, holding breath for 10 seconds, and exhaling all the gas to RV position.

(5) Six-minute walk test: The enrolled patients were performed on a flat, straight corridor with a length of 30 meters. They avoided strenuous activities within 2 hours before the test and could carry a cane or walking aid to the test. Blood pressure, pulse, and oxygen saturation were measured. Then the subjects were asked to walk as much as possible along the established route within six minutes. If they felt tired, they could slow down or rest in place and continue walking as soon as possible. At the end of the six minutes, the subjects were allowed to stay in place, and their blood pressure, pulse, and oxygen saturation were rapidly measured again, and their total distance walked was recorded.

Objects and methods of intervention According to the results of pulmonary function test, patients diagnosed as early COPD or pre-COPD were given triple bronchial inhalation therapy according to the principle of voluntary, and professional staff were arranged to explain relevant knowledge, answer questions and guide medication. Each patient was asked to record medication use.

Follow-up time and endpoint indicators The patients were followed up for 1 year from the date of enrollment. The clinical symptoms, pulmonary function parameters, and imaging parameters of early COPD and pre-COPD patients with or without triple bronchial inhalation drug use were recorded, focusing on the annual decline in FEV1% pred, FEV1/FVC and DLCO.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-70 years old; 2. smoking history ≥10 pack-years or presence of visually visible emphysema on low-dose CT scan; 3. Able to tolerate or cooperate with pulmonary function test; ④4.able to understand the study and sign the relevant informed consent.

Exclusion Criteria:

1.History of acute or chronic respiratory diseases other than COPD, including interstitial lung disease, bronchiectasis, pulmonary infection, tumor, or lung surgery; 2.patients previously diagnosed with clinical COPD; 3.Severe liver and kidney dysfunction; 4.serious heart failure or malignant arrhythmia; 5.acute cerebrovascular events within the past 3 months; 6.malignant tumor without cure; 7.the history of mental illness; 8.breastfeeding, pregnancy or planned pregnancy; 9.Subjects who are expected to be unable to cooperate and follow up.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: early chronic obstructive pulmonary disease: age < 50 years of age with at least 10 pack-years of smoking history and one of the following: FEV1/FVC< 0.7, abnormal computer tomography (CT) and a decline in FEV1 of at least 60mL/ year. Precopd (emphysema type) : Involves individuals of any age who have respiratory symptoms, with or without structural (radiographic emphysema) and/or functional abnormalities, no airflow limitation (FEV1/FVC≥0.70), and may develop persistent airflow limitation over time.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
FEV1% and FEV1/FVC | 1 year
  After one year of follow-up, FEV1% and FEV1/FVC, DLco and other indicators were observed to decrease

IPD SHARING:
Plan to Share IPD: No